CLINICAL TRIAL: NCT02845947
Title: Music Therapy During Pediatric Extubation Readiness Trials: A Pilot Study
Brief Title: Music Therapy During Pediatric Extubation Readiness Trials
Acronym: MTPERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Shawna N. Vernisie, Licensed Creative Arts Therapist - Music Therapist, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS16-0478
Record Dates: First submitted 2016-07-18; First posted 2016-07-27 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music Therapy (Experimental): Music Therapy to be provided for pediatric patients undergoing extubation readiness trial
  Interventions: Behavioral: Music Therapy
- Control (No Intervention): Patients undergoing standard extubation readiness trial

INTERVENTIONS:
Behavioral: Music Therapy — The music therapy intervention offered during the time of the patient's extubation readiness trial (ERT) will consist of live music using a multitude of instruments and patient-preferred and improvised music. The music therapy interventions will always include the use of live music, including guitar, keyboard, voice, ocean drum, reverie harp, and/or various percussive instruments. The music therapist will use a tablet to understand how to play patient-preferred songs. To ensure patient safety, the music therapist will adhere to the infection control policies set forth by the institution. The following are the intended goals of the Music therapy intervention: facilitating relaxation, alleviation of anxiety, and successful utilization of new coping skills.
  Arms: Music Therapy

SUMMARY:
This study seeks to research the effects of music therapy during pediatric extubation readiness trials. Amount of sedation, physiological measures, and parent/staff satisfaction surveys will be measured.

DETAILED DESCRIPTION:
The music therapy intervention offered during the time of the patient's extubation readiness trial (ERT) will consist of live music using a multitude of instruments and patient-preferred and improvised music. The start time and duration of the session will be initiated by the attending physician, and the length of music therapy intervention provided will not exceed two and a half hours. The music therapy intervention will continue for 30 minutes post extubation. This time frame was determined in accordance with the institution's weaning trial protocol. Family members involved in the trial, as well as the nurse and physician, will complete a post-procedural survey about the music therapy intervention.

The music therapy interventions will always include the use of live music, including guitar, keyboard, voice, ocean drum, reverie harp, and/or various percussive instruments. The music therapist will use a tablet to understand how to play patient-preferred songs. To ensure patient safety, the music therapist will adhere to the infection control policies set forth by the institution. The following are the intended goals of the Music therapy intervention: facilitating relaxation, alleviation of anxiety, and successful utilization of new coping skills.

Before the weaning trial, the music therapist will meet with the patient's family to obtain the musical preferences of the patient. During the two hour ERT, the music therapist will play patient-preferred songs on a variety of different instruments to bring about a sense of interpersonal connectedness, normalization, and to enhance adaptive coping. In order to maximize coping and minimize stress/anxiety, the music therapy intervention will be malleable and patient/family centered, responding to the changing needs that present throughout the procedure/weaning process. If the patient becomes more alert throughout the weaning process, the music therapist will adapt the music making based on patient's preferences; at this time, the patient may be able to answer yes/no questions when asked. The music therapist will adjust the volume, timbre, and tempo of the music according to the patient's respiratory rhythms throughout the weaning process and after extubation.

When the live music therapy intervention has completed, the music therapist will follow up with the family members immediately. The investigator will administer and collect the survey from the family, and the music therapist will administer and collect the survey from the nurse and physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients 0-18 years of age admitted to the pediatric intensive care unit, regardless of cognitive status
* Patients admitted receiving endotracheal mechanical ventilation

Exclusion Criteria:

* Patients receiving extubation for withdrawal of care, patients with known/documented hearing loss/deafness.
* Patients on mechanical ventilation not scheduled for planned ERT.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Music Therapy will aid in the success of extubation readiness trials as measured by physiological measures. | Through study completion, an average of 1 year.
  A data collection tool (created by the PI's) will be used to record physiological signs (heart rate and blood pressure) by a Registered Nurse (RN) every 15 minutes. The heart rate will be captured from an Intensive Care Unit monitor and the blood pressure will be measured by a blood pressure cuff administered by a RN.
Music Therapy will aid in the success of extubation readiness trials as measured by sedation bolus requirements. | Through study completion, an average of 1 year.
  A data collection tool (created by the PI's) will be used to record sedation bolus requirements (mcg/kg) every 15 minutes throughout the length of the extubation readiness trial. This will be administered and recorded by an RN.
Music Therapy will aid in the success of extubation readiness trials as measured by agitation levels. | Through study completion, an average of 1 year.
  A data collection tool (created by the PI's) will be used to record agitation levels (using the State Behavioral Scale for Mechanically Ventilated Patients) every 15 minutes throughout the length of the extubation readiness trial.
Music Therapy will reduce anxiety of physicians and nurses during the extubation readiness trial. | Through study completion, an average of 1 year.
  A survey (authored by the PI's) will be provided to physicians and nurses rating their anxiety score based on a 5-point Likert scale.
Music Therapy will reduce anxiety of parents/guardiansduring the extubation readiness trial. | Through study completion, an average of 1 year.
  A survey (authored by the PI's) will be provided to parents/guardians rating their anxiety score based on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Shawna N Vernisie, MA, Principal Investigator — Northwell Health; James B Schneider, MD, Principal Investigator — Intensivist; Mary Schafer, BSN, Principal Investigator — Northwell Health; Peter Silver, MD, Principal Investigator — Northwell Health
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradt J, Dileo C. Music interventions for mechanically ventilated patients. Cochrane Database Syst Rev. 2014;2014(12):CD006902. doi: 10.1002/14651858.CD006902.pub3. Epub 2014 Dec 9. PMID 25490233
- [Background] Thomas LA. Clinical management of stressors perceived by patients on mechanical ventilation. AACN Clin Issues. 2003 Feb;14(1):73-81. doi: 10.1097/00044067-200302000-00009. PMID 12574705
- [Background] Wong HL, Lopez-Nahas V, Molassiotis A. Effects of music therapy on anxiety in ventilator-dependent patients. Heart Lung. 2001 Sep-Oct;30(5):376-87. doi: 10.1067/mhl.2001.118302. PMID 11604980
- [Background] Chlan LL. Description of anxiety levels by individual differences and clinical factors in patients receiving mechanical ventilatory support. Heart Lung. 2003 Jul-Aug;32(4):275-82. doi: 10.1016/s0147-9563(03)00096-7. PMID 12891169
- [Background] Chlan LL. Relationship between two anxiety instruments in patients receiving mechanical ventilatory support. J Adv Nurs. 2004 Dec;48(5):493-9. doi: 10.1111/j.1365-2648.2004.03231.x. PMID 15533087
- [Background] Lee OK, Chung YF, Chan MF, Chan WM. Music and its effect on the physiological responses and anxiety levels of patients receiving mechanical ventilation: a pilot study. J Clin Nurs. 2005 May;14(5):609-20. doi: 10.1111/j.1365-2702.2004.01103.x. PMID 15840076
- [Background] Chlan L, Savik K. Patterns of anxiety in critically ill patients receiving mechanical ventilatory support. Nurs Res. 2011 May-Jun;60(3 Suppl):S50-7. doi: 10.1097/NNR.0b013e318216009c. PMID 21543962
- [Background] Li DT, Puntillo K. A pilot study on coexisting symptoms in intensive care patients. Appl Nurs Res. 2006 Nov;19(4):216-9. doi: 10.1016/j.apnr.2006.01.003. PMID 17098160
- [Background] Hofhuis JG, Spronk PE, van Stel HF, Schrijvers AJ, Rommes JH, Bakker J. Experiences of critically ill patients in the ICU. Intensive Crit Care Nurs. 2008 Oct;24(5):300-13. doi: 10.1016/j.iccn.2008.03.004. Epub 2008 May 9. PMID 18472265
- [Background] Gabor JY, Cooper AB, Crombach SA, Lee B, Kadikar N, Bettger HE, Hanly PJ. Contribution of the intensive care unit environment to sleep disruption in mechanically ventilated patients and healthy subjects. Am J Respir Crit Care Med. 2003 Mar 1;167(5):708-15. doi: 10.1164/rccm.2201090. PMID 12598213
- [Background] Chlan L. A review of the evidence for music intervention to manage anxiety in critically ill patients receiving mechanical ventilatory support. Arch Psychiatr Nurs. 2009 Apr;23(2):177-9. doi: 10.1016/j.apnu.2008.12.005. PMID 19327560
- [Background] Hunter BC, Oliva R, Sahler OJ, Gaisser D, Salipante DM, Arezina CH. Music therapy as an adjunctive treatment in the management of stress for patients being weaned from mechanical ventilation. J Music Ther. 2010 Fall;47(3):198-219. doi: 10.1093/jmt/47.3.198. PMID 21275332
- [Background] Korhan EA, Khorshid L, Uyar M. The effect of music therapy on physiological signs of anxiety in patients receiving mechanical ventilatory support. J Clin Nurs. 2011 Apr;20(7-8):1026-34. doi: 10.1111/j.1365-2702.2010.03434.x. Epub 2011 Feb 16. PMID 21323778
- [Background] Hetland B, Lindquist R, Chlan LL. The influence of music during mechanical ventilation and weaning from mechanical ventilation: A review. Heart Lung. 2015 Sep-Oct;44(5):416-25. doi: 10.1016/j.hrtlng.2015.06.010. Epub 2015 Jul 27. PMID 26227333
- [Background] Johnson MM, Sexton DL. Distress during mechanical ventilation: patients' perceptions. Crit Care Nurse. 1990 Jul-Aug;10(7):48-57. No abstract available. PMID 2403412
- [Background] Loomba RS, Arora R, Shah PH, Chandrasekar S, Molnar J. Effects of music on systolic blood pressure, diastolic blood pressure, and heart rate: a meta-analysis. Indian Heart J. 2012 May-Jun;64(3):309-13. doi: 10.1016/S0019-4832(12)60094-7. PMID 22664817
- [Background] Tracy MF, Chlan L. Nonpharmacological interventions to manage common symptoms in patients receiving mechanical ventilation. Crit Care Nurse. 2011 Jun;31(3):19-28. doi: 10.4037/ccn2011653. PMID 21632591
- [Background] Chlan LL, Weinert CR, Heiderscheit A, Tracy MF, Skaar DJ, Guttormson JL, Savik K. Effects of patient-directed music intervention on anxiety and sedative exposure in critically ill patients receiving mechanical ventilatory support: a randomized clinical trial. JAMA. 2013 Jun 12;309(22):2335-44. doi: 10.1001/jama.2013.5670. PMID 23689789
- [Background] Davis T, Jones P. Music therapy: decreasing anxiety in the ventilated patient: a review of the literature. Dimens Crit Care Nurs. 2012 May-Jun;31(3):159-66. doi: 10.1097/DCC.0b013e31824dffc6. PMID 22475701
- [Background] Azoulay E, Chaize M, Kentish-Barnes N. Involvement of ICU families in decisions: fine-tuning the partnership. Ann Intensive Care. 2014 Nov 30;4:37. doi: 10.1186/s13613-014-0037-5. eCollection 2014. PMID 25593753